CLINICAL TRIAL: NCT05862766
Title: A Pilot Study of Isatuximab in Addition to Standard Therapy for Desensitization or Antibody-mediated Rejection in Lung Transplant Recipients
Brief Title: Isatuximab in Lung Transplant Recipients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study no longer had funding and therefore was closed before enrollment began.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-00992
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Antibody-mediated Rejection; Allosensitization
Keywords: Desensitization; antibody-mediated rejection; isatuximab
MeSH Terms: interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Peri-transplant desensitization group (Experimental): Listed and will receive a lung transplant or multi-organ transplant involving a lung at NYU Langone Health that is deemed to require peri-transplant desensitization. Participants will be treated with standard-of-care consisting of plasmaspheresis, IVIG, rituximab and the experimental agent, isatuximab. Patients will be followed with standard-of-care immunologic assessment consisting of weekly DSA assessment and flow cytometry crossmatch (only in the desensitization arm). Additionally, participants will have a bone marrow biopsy with pathologic examination and cell counts performed at the time of transplant and repeated at the 30-day bronchoscopy to assess for plasma cell elimination
  Interventions: Drug: Isatuximab; Procedure: bone marrow biopsy
- Treatment of antibody-mediated rejection (Experimental): Received a lung transplant or multi-organ transplant involving a lung at NYU Langone Health. Participants will be treated with standard-of-care consisting of plasmaspheresis, IVIG, rituximab and the experimental agent, isatuximab.
  Interventions: Drug: Isatuximab

INTERVENTIONS:
Drug: Isatuximab — The dose will consist of isatuximab 10 mg/kg actual body weight given weekly for the first 4 weeks, followed by 10 mg/kg biweekly for an additional 4 doses. Isatuximab is a clear, colorless to slightly yellow solution. It is supplied as 100 mg/5 mL or 500 mg/25 mL single-dose vials.
  Other Names: SARCLISA®
Procedure: bone marrow biopsy — Bone marrow biopsy at the time of lung transplantation and at approximately 1 month following completion of therapy. Initial bone marrow biopsy to be performed during the lung transplant operation and to be collected from the sternum by the operating surgeon. Follow-up bone marrow biopsy to be completed by credentialed hematologist during a regularly scheduled follow-up bronchoscopy with standard procedural anesthesia sedation.
  Arms: Peri-transplant desensitization group

SUMMARY:
The purpose of this study is to determine the safety and feasibility of adding isatuximab to standard of care therapies in patients who will receive a lung transplant, but have significant antibodies against the donor (desensitization), or patients who have previously received a lung transplant and develop antibodies against the donor (antibody-mediated rejection, AMR). The study will compare the impact of isatuximab on the recurrence of antibodies after they have been removed from the blood by a process known as plasmapheresis that is standard of care for this condition. The use of isatuximab in lung transplant recipients is investigational, meaning it is not Food and Drug Administration (FDA) approved for use in lung transplant recipients. This study is a pilot study investigating the feasibility and safety of isatuximab in lung transplant patients. Isatuximab is an FDA approved drug indicated for the treatment of multiple myeloma. It may also be useful for transplant recipients with antibodies against the donor because it eliminates the cells that make antibodies.

DETAILED DESCRIPTION:
This dual-arm pilot study will enroll approximately 6 patients undergoing lung transplantation at NYU Langone Health who are either receiving peri-transplant desensitization, or who are admitted for treatment of AMR. All patients will be treated with standard-of-care consisting of plasmaspheresis, IVIG, and rituximab. Additionally, the experimental agent, isatuximab, will be added to this treatment protocol. The patients will first receive 4 weekly doses of isatuximab, followed by 4 bi¬-weekly doses (total 8 doses given over 12 weeks). Patients will be followed with standard-of-care immunologic assessment consisting of weekly DSA assessment and flow cytometry crossmatch (only in the desensitization arm). Additionally, patients undergoing peri-transplant desensitization will have a bone marrow biopsy with pathologic examination and cell counts performed at the time of transplant and repeated at the 30-day bronchoscopy to assess for plasma cell elimination.

ELIGIBILITY:
Inclusion Criteria:

Cohort A (Desensitization) Inclusion Criteria:

* Age ≥ 18 years
* Listed and will receive a lung transplant or multi-organ transplant involving a lung at NYU Langone Health that is deemed to require peri-transplant desensitization
* Able and willing to provide informed consent
* Pre-transplant DSA > 5,000 MFI in undiluted serum (measured as individual DSA MFI or as sum of multiple DSAs >1000 MFI in the undiluted serum)

Cohort B (AMR) Inclusion Criteria:

* Age ≥ 18 years
* Received a lung transplant or multi-organ transplant involving a lung at NYU Langone Health
* Able and willing to provide informed consent
* Allograft dysfunction in the setting of at least one of the following criteria:
* Histopathology suggestive of AMR
* Lung biopsy demonstrating C4d deposition
* Positive DSA > 2,000 MFI (as individual DSA MFI)

Exclusion Criteria:

* Prior or current treatment with rituximab within 6 months of isatuximab administration
* Prior or current treatment with tocilizumab within 6 months of isatuximab administration
* Contraindication to isatuximab due to intolerance or hypersensitivity
* Pregnant or breastfeeding women
* Known malignancy
* Active infection without adequate treatment or source control
* Known hepatitis B viral infection
* Known HIV infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Resolution, as measured by the number of participants with less than 1 episode of Antibody-mediated rejection (AMR) | Day 0 (Visit 1)
  Participants undergoing desensitization will have stable supplemental oxygen requirement or no supplemental oxygen requirement
Clinical Resolution, as measured by the number of participants with less than 1 episode of Antibody-mediated rejection (AMR) | Day 28 (Visit 5)
  Participants undergoing desensitization will have stable supplemental oxygen requirement or no supplemental oxygen requirement
Clinical Resolution, as measured by the number of participants with no presence of Donor-specific antibody (DSA) | Day 0 (Visit 1)
  Participants undergoing desensitization will have no presence of Donor-specific-antibody
Clinical Resolution, as measured by the number of participants with no presence of Donor-specific antibody (DSA) | Day 28 (Visit 5)
  Participants undergoing desensitization will have no presence of Donor-specific-antibody
Clinical Resolution, as measured by the number of participants with reduction of DSA titer | Day 0 (Visit 1)
  Participants undergoing desensitization will have no presence of Donor-specific-antibody measured by DSA titer or by C1q assay.
Clinical Resolution, as measured by the number of participants with reduction of DSA titer | Day 28 (Visit 5)
  Participants undergoing desensitization will have no presence of Donor-specific-antibody measured by DSA titer or by C1q assay.

SECONDARY OUTCOMES:
Change in effects of pre-treatment Donor-Specific-Antibodies (DSAs ) with <2000 Mean fluorescent intensity (MFI) at 1:16 dilution | Day 0 (Visit 1), Day 14 (Visit 3), Day 28 (Visit 5), Day 56 (Visit 7), Day 84 (Visit 9)
  Percent Mean fluorescent intensity (MFI) change in undiluted serum
Change in effects of pre-treatment Donor-Specific-Antibodies (DSAs ) with 2001-7999 Mean fluorescent intensity (MFI) at 1:16 dilution | Day 0 (Visit 1), Day 14 (Visit 3), Day 28 (Visit 5), Day 56 (Visit 7), Day 84 (Visit 9)
  Percent moderate titer DSA with <1000 Mean fluorescent intensity (MFI) at 1:16 dilution
Change in effects of pre-treatment Donor-Specific-Antibodies (DSAs ) ≥ 8000 Mean fluorescent intensity (MFI) at 1:16 dilution | Day 0 (Visit 1), Day 14 (Visit 3), Day 28 (Visit 5), Day 56 (Visit 7), Day 84 (Visit 9)
  Percent Mean fluorescent intensity (MFI) reduction of high titer DSAs at 1:16 dilution

CONTACTS AND LOCATIONS:
Overall Officials: Luis Angel, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request and as agreed upon by the study team members.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to tyler.lewis@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.